CLINICAL TRIAL: NCT01309594
Title: A Safety and Efficacy Study of Autologous Bone Marrow Cell Infusion Therapy in HIV Infected Patients With Advanced Liver Cirrhosis
Brief Title: HIV Liver Regeneration Project for HIV Patients With Cirrhosis by Autologous Bone Marrow Transplantation
Acronym: HIV-ABMi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Center for Global Health and Medicine, Japan (Other Government)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWA00005823-AMBi2011; UMIN000005174 (Other: University Hospital Medical Information Network (UMIN))
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infection; AIDS; Cirrhosis
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Fibrosis | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic stem cell transplantation (Experimental): Extraction of bone marrow cells from HIV positive patients with advanced liver cirrhosis and transplant their bone marrow back into the patients
  Interventions: Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — Harvest and apheresis of bone marrow cells from HIV infected patients with cirrhosis under general anesthesia, using bone marrow collection system and transplanting the patients' hematopoietic stem cells back to the patients
  Other Names: Autologous bone marrow cell infusion therapy (ABMi)

SUMMARY:
An international investigation to evaluate if, and if so how long, autologous bone marrow hematopoietic stem cell transplantation can safely restore liver functions for HIV infected patients who have decompensated liver cirrhosis.

DETAILED DESCRIPTION:
An international investigation to evaluate if, and if so how long, autologous bone marrow (ABM) hematopoietic stem cell transplantation (HSCT) can safely restore liver functions for HIV infected patients who have decompensated liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria: Outpatients or inpatients that are treated for HIV infection at AIDS Clinical Center of National Center for Global Health and Medicine who meet all criteria following:

* have cirrhosis with 7 or higher Child-Pugh Score in Child-Pugh Score B
* able to consent and willing to participate in the study
* under good control for HIV infection

Exclusion Criteria: Cases applicable to ANY condition of the following:

* Hepatocellular carcinoma (HCC), except for cases having been completely treated without history of recurrence
* Malignant tumors other than HCC
* Alcoholic liver disease (ALD)
* Hemoglobin under 8g/dL or Platelets under 20/ml at the registration
* Esophageal or gastric varices with a risk of bursting, except for cases with only cured history of such conditions
* Cases that cannot obtain the informed consent to autologous blood transfusion
* Pregnancy
* Renal dysfunction with 2mg/dL or higher serum creatinine
* Performance Status 3 or 4 (assessment excludes hemophilic arthritis related daily life limitations)
* Cases not fit for general anesthesia
* Other conditions considered not suitable for the study by doctors

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Post-transplantation prognosis for cirrhosis | 24 weeks
  Evaluate statistical significance between pre-transplantation and 24 weeks after in:
  * Child-Pugh score
  * albumin
  * serum fibrosis markers
  * Transient Elastography (TM)
  * ascites imagery
  * SF-36v2(TM) Health Survey.
  Because advanced liver cirrhosis is a progressive condition itself, treatment efficacy is defined by "improvement" and "no change" in the indicators listed.

SECONDARY OUTCOMES:
Duration of the treatment efficacy | After 24 weeks up to 48 weeks
  Using the same evaluation modules as of the primary outcomes, investigate and assess the autologous bone marrow transplantation effectivity chronologically after the primal 24 weeks up to 48 weeks to evaluate the duration of the treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Oka, MD PhD, Principal Investigator — National Center for Global Health and Medicine
Locations (1):
- National Center for Global Health and Medicine, Shinjuku, Tokyo, Japan